CLINICAL TRIAL: NCT03904277
Title: Does Patent Foramen Ovale Size Matter in Men and Women
Status: Completed | Type: Observational
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Other Study IDs: 04302018.049
Record Dates: First submitted 2019-04-01; First posted 2019-04-05 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-09

CONDITIONS: Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma from venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No PFO: Research subjects who present no evidence of PFO - IE no appearance of saline contrast microbubbles within 3 cardiac cycles
- Small PFO: Research subjects who present evidence of having a small PFO or ASD - IE appearance of 1-11 saline contrast microbubbles within 3 cardiac cycles
- Large PFO: Research subjects who present evidence of having a large PFO - IE appearance of 12+ saline contrast microbubbles within 3 cardiac cycles.

SUMMARY:
A patent foramen ovale (PFO) is present in ~30% of the general population. The PFO has historically been considered to be trivial. However, recent work by the investigator's group and others has identified that, compared to individuals without a PFO, those with a PFO have worse pulmonary gas exchange efficiency, have a higher core body temperature, blunted ventilatory responses to chronic hypoxia and acute carbon dioxide and increased susceptibility to altitude illnesses such as acute mountain sickness, and high altitude pulmonary edema (Lovering, Elliott & Davis J Appl Physiol 2016). Specific to this application,subjects with a PFO may have worse pulmonary gas exchange efficiency because a PFO is a potential source of right-to-left shunt that will make pulmonary gas exchange efficiency worse. If true, then this may negatively impact exercise capacity and/or exercise tolerance. Further, in those with a PFO compared to those without, preliminary work from the investigator's lab indicates that there may be an effect of PFO size on pulmonary gas exchange efficiency. This is such that those with a large PFO (grade 3 or higher) display significantly worse gas exchange efficiency compared to those with a small (grade 2 or lower) or no PFO,even at low exercise workloads. Additionally, the investigators were curious as to whether there would be a sex effect, but due to logistical constraints, the investigators were unable to recruit an equal number of female and male subjects. Thus, in addition to the potential size effect on the investigators outcome measures, the investigators would like to build on this work by examining the potential effect of biological sex. Although a PFO has been traditionally considered to have a minimal impact of physiology and pathophysiology, emerging evidence suggests this may not be the case. The investigator's lab is focused on understanding how and why a relatively small hole in the heart (PFO) can have a relatively large impact on cardiopulmonary and respiratory physiology, and how these impacts may be based on the size of the PFO.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-40
* Known to have/not have a PFO.

Exclusion Criteria:

* Previous history of coronary artery disease(ischemic heart disease such as angina, heart attack, myocardial infarction).
* Failure of Modified Allen's Test in both hands.
* Currently taking medications or herbal supplements for any heart or respiratory disease that they cannot stop taking for 48 hrsprior to testing (seasonal allergy medication not included in exclusion medications).
* Lidocaine, nitroglycerine or heparin allergy.
* Women who are pregnant or trying to become pregnant.
* Previous history of any condition that would prevent the subject from performing cycle ergometer exercise (for exercise study only).

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Healthy adults aged 18-40 with and without a PFO.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
alveolar-arterial difference in oxygen | Baseline
  difference in the partial pressure of oxygen between the alveoli (calculated) and arterial blood (direct measure)
aerobic exercise capacity | Baseline
  ability to utilize oxygen while exercising, AKA Vo2MAX
six-minute walk test | Baseline
  distance covered in 6 minutes of walking
minute flow of intrapulmonary areterio-venous anastamoses (QIPAVA) | Baseline
  minute flow through intrapulmonary arteriovenous anastamoses
core body temperature | Baseline
  subject's core body temperature as measured through an ingestible pill
level of tumor necrosis factor alpha | Baseline
  inflammatory marker
level of C-C motif cytokine 2 | Baseline
  inflammatory marker
level of interferon alpha 2 | Baseline
  inflammatory marker
level of interferon gamma | Baseline
  inflammatory marker
level of interleukin 1 beta | Baseline
  inflammatory marker
level of interleukin 6 | Baseline
  inflammatory marker
level of interleukin 8 | Baseline
  inflammatory marker
level of interleukin 10 | Baseline
  inflammatory marker
level of interleukin 12p70 | Baseline
  inflammatory marker
level of interleukin 17 alpha | Baseline
  inflammatory marker
level of interleukin 18 | Baseline
  inflammatory marker
level of interleukin 23 | Baseline
  inflammatory marker
level of interleukin 33 | Baseline
  inflammatory marker
level of myoglobin | Baseline
  inflammatory marker
level of myeloid-related protein 8/14 | Baseline
  inflammatory marker
level of neutrophil gelatinase-associated lipocalin | Baseline and 3 months post percutaneous closure
  inflammatory marker
level of c-reactive protein | Baseline
  inflammatory marker
matrix metallopeptidase 2 | Baseline and 3 months post percutaneous closure
  inflammatory marker
level of osteopontin | Baseline
  inflammatory marker
level of myloperoxidase | Baseline
  inflammatory marker
level of Serum amyloid A | Baseline
  inflammatory marker
level of insulin like growth factor binding protein 4 | Baseline
  inflammatory marker
level of intracellular adhesion molecule 1 | Baseline
  inflammatory marker
level of vascular cell adhesion protein 1 | Baseline
  inflammatory marker
level of metallopeptidase 9 | Baseline
  inflammatory marker
level of Cystatin C | Baseline
  inflammatory marker

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiorespiratory and Pulmonary Physiology Lab, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT03904277/Prot_SAP_000.pdf